CLINICAL TRIAL: NCT07289282
Title: The Relationship Between microRNAs in Breast Cancer Subtypes and Response to Neoadjuvant Chemotherapy and Pathological Response
Brief Title: Circulating microRNAs and Response to Neoadjuvant Chemotherapy in Breast Cancer
Acronym: miRNA-NAC
Status: Not yet recruiting | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Emine YILDIRIM, associate professor, MD, Atlas University
Other Study IDs: Breast-miRNA
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Pathological Response; Invasive Breast Carcinoma; MicroRNAs
Keywords: microRNA; Circulating microRNAs; Neoadjuvant Chemotherapy; Pathological Complete Response; Predictive Biomarkers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Cohort

SUMMARY:
This prospective observational study aims to investigate subtype-specific circulating microRNAs (miRNAs) and their association with response to neoadjuvant chemotherapy (NAC) in patients with breast cancer. Serum samples will be collected before NAC and prior to surgery, and changes in miRNA expression levels will be evaluated. Pathological complete response (pCR) and Miller-Payne scoring will be used to assess treatment response after NAC. The study also explores whether changes in circulating miRNA profiles can predict treatment response across different breast cancer subtypes. The findings may help identify biomarkers that support treatment planning and personalized therapy strategies.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study designed to evaluate circulating microRNA (miRNA) expression patterns in breast cancer patients receiving neoadjuvant chemotherapy (NAC). The primary aim is to examine changes in selected miRNAs (including miR-200 family members, miR-34a, miR-221/222, miR-155, and miR-146a) before NAC initiation and prior to surgery, and to determine their association with pathological response.

Participants diagnosed with breast cancer and scheduled to receive standard NAC will be enrolled consecutively. Serum samples will be collected at two time points: (1) before NAC initiation, and (2) following completion of NAC but before surgery. Quantitative RT-PCR methods will be used to measure circulating miRNA expression levels. Pathological response will be evaluated using pathological complete response (pCR) status and Miller-Payne tumor regression grading.

Secondary aims include examining the relationship between miRNA dynamics and breast cancer subtypes, evaluating the potential predictive value of miRNAs for NAC response, and assessing possible correlations between circulating tumor cell (CTC) levels and treatment outcomes. No investigational drugs or devices will be used in this study, and all treatments will follow standard clinical protocols.

The study is expected to contribute to the identification of minimally invasive biomarkers that may support personalized treatment approaches and improve prediction of NAC response in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* Planned to receive neoadjuvant chemotherapy
* Biologically female
* Age ≥ 18 years
* Ability to provide informed consent
* Adequate organ function to receive standard NAC (based on routine clinical evaluation)

Exclusion Criteria:

* Presence of metastatic disease at diagnosis
* Prior systemic chemotherapy for breast cancer
* Pregnancy or breastfeeding
* Active infection or uncontrolled comorbid conditions interfering with study participation
* Any condition preventing collection of blood samples

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with breast cancer who are scheduled to undergo standard neoadjuvant chemotherapy at a single tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in circulating microRNA expression levels before and after neoadjuvant chemotherapy | Baseline (before NAC) and pre-surgery (after completion of NAC)
  Quantitative assessment of selected serum microRNAs (miR-200a/b/c, miR-34a, miR-221/222, miR-155, miR-146a) using RT-PCR. Changes in expression levels will be compared between baseline and pre-surgery samples.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Yildirim, MD, Principal Investigator — Atlas University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and data protection regulations. Only de-identified aggregated results may be shared upon reasonable request.